CLINICAL TRIAL: NCT03652532
Title: Effects of Alternate Day Fasting and Exercise on Body Weight, Visceral Fat, and Metabolic Parameters in Overweight or Obese Adults: A Randomized Controlled Trial
Brief Title: Alternate Day Fasting and Exercise in Overweight or Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-Won Lee, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2014-0117
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Overweight; Obesity; Diet Modification; Exercise
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alternate Day Fasting and Exercise (Experimental)
  Interventions: Behavioral: Alternate Day Fasting; Behavioral: Exercise
- Alternate Day Fasting (Experimental)
  Interventions: Behavioral: Alternate Day Fasting
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Control (No Intervention): regular eating and exercise habits for 8 weeks

INTERVENTIONS:
Behavioral: Alternate Day Fasting — During the 8-week intervention, participants consumed 25% of their daily recommended energy intake (approximately 500 kcal) on each "fast day" (24 h), and consumed food ad libitum on each "feed day" (24 h). The "fast day" and "feed day" were repeated every other day, and the "fast day" occurred 3 days per week.
  Arms: Alternate Day Fasting; Alternate Day Fasting and Exercise
Behavioral: Exercise — During the 8-week intervention, participants visited the research center gym at least three times per week and received exercise logs. Each exercise session began with 5 minutes of warm-up and ended with 5 minutes of cool-down. Resistance training was performed using weight training machines, barbells, and dumbbells for 40 minutes. Aerobic exercise was performed on motorized treadmills for 20 minutes.
  Arms: Alternate Day Fasting and Exercise; Exercise

SUMMARY:
Alternate day fasting is known to be helpful to control weight and have a positive effect on insulin resistance and cardiovascular risk factors. However, there have been no studies on weight reduction program combining alternate day fasting with exercise which preserves lean mass in Korea. The purpose of this randomized clinical trial is to examine the effects of alternate day fasting and exercise on weight reduction, visceral fat, and metabolic parameters in overweight or obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-65 years
* Body mass index (BMI) more than 23.0 kg/m² (overweight or obese for Asian populations, according to the World Health Organization)

Exclusion Criteria:

* Participants with weight gain more than 5kg in the last 3 months
* Participants with history of bariatric surgery
* Participants with secondary obesity, such as hypothyroidism
* Participants with uncontrolled hypertension or type 1 diabetes
* Participants who are taking anti-diabetic medications due to type 2 diabetes
* Participants with hepatic disease (AST or ALT ≥200 mg/dL)
* Participants with renal disease (serum creatinine ≥2.0 mg/dL)
* Participants with pancreatitis or related disorders
* Participants with acute infectious diseases (i.e., pneumonia, acute enteritis, or urinary infection)
* Participants with chronic inflammatory diseases (i.e., rheumatoid arthritis, or lupus)
* Participants with overeating behavior
* Participants with history of cardiovascular diseases
* Participants with history of cancer
* Participants who are taking anti-obesity, anti-diabetic, diuretic, central-nervous system, antidepressant, antipsychotic, or steroid medications
* Pregnant or lactating women
* Participants who intake more than 30 g of alcohol daily
* Night-time or shift-work workers
* Participants with chronic malabsorption syndrome or cholestasis
* Participants with other medical conditions that would preclude subjects from participating in exercise and physical test

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2016-03-08 (Actual); Study Completion 2016-03-08 (Actual)

PRIMARY OUTCOMES:
Change in body weight | baseline, 8 weeks
  body weight (kg)

SECONDARY OUTCOMES:
Change in visceral fat | baseline, 8 weeks
  visceral fat areas (cm2) measured by fat measurement computed tomography (CT)
Change in fasting glucose | baseline, 8 weeks
  fasting glucose (mg/dL)
Change in insulin | baseline, 8 weeks
  insulin (mcIU/mL)
Change in triglyceride | baseline, 8 weeks
  triglyceride (mg/dL)
Change in high-density lipoprotein cholesterol (HDL-cholesterol) | baseline, 8 weeks
  HDL-cholesterol (mg/dL)
Change in low-density lipoprotein cholesterol (LDL-cholesterol) | baseline, 8 weeks
  LDL-cholesterol (mg/dL) calculated using the Friedewald equation

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Oh M, Kim S, An KY, Min J, Yang HI, Lee J, Lee MK, Kim DI, Lee HS, Lee JW, Jeon JY. Effects of alternate day calorie restriction and exercise on cardio-metabolic risk factors in overweight and obese adults: an exploratory randomized controlled study. BMC Public Health. 2018 Sep 15;18(1):1124. doi: 10.1186/s12889-018-6009-1. PMID 30219052